CLINICAL TRIAL: NCT05019976
Title: An i3+3 Phase I Dose-per-Fraction Escalation Trial for Relapsed/Refractory Hodgkin/Non-Hodgkin Lymphoma
Brief Title: Radiation Dose Study for Relapsed/Refractory Hodgkin/Non-Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB21-0666
Record Dates: First submitted 2021-08-20; First posted 2021-08-25 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Non-hodgkin Lymphoma; Hodgkin Lymphoma; Lymphoma
Keywords: cancer; lymph nodes; cancer in lymph nodes
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Dose-Finding Group 0 - Dose Level 0 (Experimental): High-energy radiation will be delivered to a focused area of your body using a treatment machine called a linear accelerator. Radiation will be delivered through an IV. A mold will also be customized to fit your body, so you don't move during the radiation process. The actual time on the radiation treatment machine will be 30-60 minutes. The mold will be removed after the treatment.
  The longest possible treatment will be 14 radiation treatments over a course of 3 weeks. The shortest possible treatment will be 3 treatments in duration or less than 1 week. The amount of time required for radiation treatment depends on the dose group your are assigned.
  Participants will receive radiation to at least 1 but no more than 5 lesions (areas of body with cancer).
  Interventions: Radiation: Radiation - Dose Level 0
- Dose-Finding Group 1 - Dose Level 1 (Experimental): High-energy radiation will be delivered to a focused area of your body using a treatment machine called a linear accelerator. Radiation will be delivered through an IV. A mold will also be customized to fit your body, so you don't move during the radiation process. The actual time on the radiation treatment machine will be 30-60 minutes. The mold will be removed after the treatment.
  The longest possible treatment will be 14 radiation treatments over a course of 3 weeks. The shortest possible treatment will be 3 treatments in duration or less than 1 week. The amount of time required for radiation treatment depends on the dose group your are assigned.
  Participants will receive radiation to at least 1 but no more than 5 lesions (areas of body with cancer).
  Interventions: Radiation: Radiation - Dose Level 1
- Dose-Finding Group 2 - Dose Level 2 (Experimental): High-energy radiation will be delivered to a focused area of your body using a treatment machine called a linear accelerator. Radiation will be delivered through an IV. A mold will also be customized to fit your body, so you don't move during the radiation process. The actual time on the radiation treatment machine will be 30-60 minutes. The mold will be removed after the treatment.
  The longest possible treatment will be 14 radiation treatments over a course of 3 weeks. The shortest possible treatment will be 3 treatments in duration or less than 1 week. The amount of time required for radiation treatment depends on the dose group your are assigned.
  Participants will receive radiation to at least 1 but no more than 5 lesions (areas of body with cancer).
  Interventions: Radiation: Radiation - Dose Level 2
- Dose-Finding Group 3 - Dose Level 3 (Experimental): High-energy radiation will be delivered to a focused area of your body using a treatment machine called a linear accelerator. Radiation will be delivered through an IV. A mold will also be customized to fit your body, so you don't move during the radiation process. The actual time on the radiation treatment machine will be 30-60 minutes. The mold will be removed after the treatment.
  The longest possible treatment will be 14 radiation treatments over a course of 3 weeks. The shortest possible treatment will be 3 treatments in duration or less than 1 week. The amount of time required for radiation treatment depends on the dose group your are assigned.
  Participants will receive radiation to at least 1 but no more than 5 lesions (areas of body with cancer).
  Interventions: Radiation: Radiation - Dose Level 3
- Dose-Finding Group 4 - Dose Level 4 (Experimental): High-energy radiation will be delivered to a focused area of your body using a treatment machine called a linear accelerator. Radiation will be delivered through an IV. A mold will also be customized to fit your body, so you don't move during the radiation process. The actual time on the radiation treatment machine will be 30-60 minutes. The mold will be removed after the treatment.
  The longest possible treatment will be 14 radiation treatments over a course of 3 weeks. The shortest possible treatment will be 3 treatments in duration or less than 1 week. The amount of time required for radiation treatment depends on the dose group your are assigned.
  Participants will receive radiation to at least 1 but no more than 5 lesions (areas of body with cancer).
  Interventions: Radiation: Radiation - Dose Level 4

INTERVENTIONS:
Radiation: Radiation - Dose Level 0 — Dose Per Fraction (Each Radiation Treatment): 3.2Gy to 2.4Gy (minimal dose) depending on what study doctor prescribes
  Total Dose of Radiation for Treatment Period: 44.8Gy to 33.6Gy (minimal dose) depending on what study doctor prescribes
  Total Number of Radiation Treatments: 14
  Arms: Dose-Finding Group 0 - Dose Level 0
Radiation: Radiation - Dose Level 1 — Dose Per Fraction (Each Radiation Treatment): 4.2Gy to 3.2Gy (minimal dose) depending on what study doctor prescribes
  Total Dose of Radiation for Treatment Period: 42Gy to 32Gy (minimal dose) depending on what study doctor prescribes
  Total Number of Radiation Treatments: 10
  Arms: Dose-Finding Group 1 - Dose Level 1
Radiation: Radiation - Dose Level 2 — Dose Per Fraction (Each Radiation Treatment): 5.2Gy to 4.2Gy (minimal dose) depending on what study doctor prescribes
  Total Dose of Radiation for Treatment Period: 39.2Gy to 29.4Gy (minimal dose) depending on what study doctor prescribes
  Total Number of Radiation Treatments: 7
  Arms: Dose-Finding Group 2 - Dose Level 2
Radiation: Radiation - Dose Level 3 — Dose Per Fraction (Each Radiation Treatment): 6.8Gy to 5.4Gy (minimal dose) depending on what study doctor prescribes
  Total Dose of Radiation for Treatment Period: 34Gy to 27Gy (minimal dose) depending on what study doctor prescribes
  Total Number of Radiation Treatments: 5
  Arms: Dose-Finding Group 3 - Dose Level 3
Radiation: Radiation - Dose Level 4 — Dose Per Fraction (Each Radiation Treatment): 10Gy to 7.8Gy (minimal dose) depending on what study doctor prescribes
  Total Dose of Radiation for Treatment Period: 30Gy to 23.4Gy (minimal dose) depending on what study doctor prescribes
  Total Number of Radiation Treatments: 3
  Arms: Dose-Finding Group 4 - Dose Level 4

SUMMARY:
This study focuses on using shortened courses of radiation for participants with relapsed/refractory Hodgkin/Non-Hodgkin lymphoma. Treatment radiation over 5-6 weeks is often standard of care for many people with lymphoma, but doctors leading this study aim to find out if using radiation for a shorter period of time can be safe for treating lymphoma and if so, what is the safest shortened dose of radiation for participants.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Signed Written Informed Consent:

   * Participants must be able to give self-consent and then sign and date an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)-approved written informed consent in accordance with local regulatory and institutional guidelines. This consent must be obtained before the performance of any protocol-related procedures that are not considered part of normal participant care.
   * Participants must be willing and able to comply with scheduled visits, treatment schedule, laboratory testing, and other requirements of the study.
2. Must have the following disease/participant characteristics:

   * Men or women ≥ 18 years of age.
   * Must have clinically confirmed relapsed/refractory Hodgkin/non-Hodgkin lymphoma
   * Mush have undergone appropriate standard of care treatment options (in the opinion of the treating investigator).
   * Must have measurable disease/tumors as defined by RECIST Version 1.1, including at least one tumor lesion that meets criteria for radiation (0.25 cc to 65 cc of viable tumor approximately 5 cm in maximal dimension). Tumors larger than 65 cc can be partially treated but the whole tumor should receive at least the minimal prescribed dose.
   * Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
   * Must have adequate organ function, as defined by clinical lab values provided to the study doctor.
   * Must have an doctor-determined life expectancy of at least 1 month.
   * Participants who are women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 72 hours prior to the start of study.
   * Participants who are women must not be breastfeeding.
   * Participants who are WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) and up to 5 months post last dose of study drug(s).
   * Participants who are WOCBP who are continuously not heterosexually active are exempted from contraceptive requirements but still must undergo pregnancy testing as described in this section.
   * Participants who are males and who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) and up to 7 months post last dose of study drug(s). In addition, male participants must be willing to refrain from sperm donation during this time.
   * Participants who are azoospermic males (males who dont ejaculate without sperm) are exempt from contraceptive requirements.
   * Study doctors shall counsel WOCBP, and male participants who are sexually active with WOCBP, on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise on the use of highly effective methods of contraception, which have a failure rate of < 1% when used consistently and correctly.

EXCLUSION CRITERIA:

* Participants must not have an indolent lymphoma or other type of lymphoma which could be effectively treated with radiation doses substantially less then and EQD2 of 50 Gy
* Participants must not receive concurrent chemotherapy, targeted small molecule therapy, radiation or other anti-cancer therapy (with exceptions for disease-specific hormone treatments considered standard of care), anti-cancer monoclonal antibody (mAb) or have not recovered (i.e. < grade 1 or at baseline) from adverse events due to a previously administered agent. Participants may receive concurrent steroids.

  i) Note: subjects with < grade 2 neuropathy are an exception to this criterion and may qualify for the study.

ii) Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.

iii) Note: subjects with any grade alopecia are an exception to this criterion and may qualify for the study

* Participants must not have had prior radiation therapy (defined as >10% of prior prescription dose) to the area planning to be treated with radiation.
* Participants who have had prior cytotoxic chemotherapy must not receive that therapy within 2 weeks of the initiation of radiation
* Participants who have had prior anti-cancer monoclonal antibody (mAb) or other small molecules must not receive that therapy within 7 days of the initiation of radiation
* Participants must not have a known additional malignancy that could confuse analysis of on-study treatment. Inclusion of all study participants with more than one malignancy must be discussed and approved by the PI.
* Participants must not have a known history of non-infectious pneumonitis that required steroids for treatment.
* Participants must not have evidence of interstitial lung disease.
* Participants must not have a current seizure disorder.
* Participants must not have a history or current evidence of any condition, therapy or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
* If known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected) then patient is not eligible for treatment of liver lesions
* Participants must not have had uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:

  * Myocardial infarction or stroke/transient ischemic attack within the past 6 months
  * Uncontrolled angina within the past 3 months
  * Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
  * History of other clinically significant heart disease (e.g. cardiomyopathy, congestive heart failure with New York Heart Association functional classification III to IV, pericarditis, significant pericardial effusion, or myocarditis)
  * Cardiovascular disease-related requirement for daily supplemental oxygen therapy.
* Participants may not concomitantly use statins while on study. However, a patient using statins for over 3 months prior to study drug administration and in stable status without CK rise may be permitted to enroll.
* Participants may not have current or history of clinically significant muscle disorders (e.g. myositis), recent unresolved muscle injury, or any condition known to elevate serum CK levels.
* Participants must not be prisoners or be involuntarily incarcerated.
* Participants must not be compulsorily detained for treatment of either a psychiatric or physical (e.g., infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose Per Fraction of Radiation | 1 Month
  Maximum tolerated dose of radiation per fraction among participants with relapsed/refractory Hodgkin/non-Hodgkin lymphoma as assessed by dose-limiting toxicities (severe side effects that limit the dose of radiation) defined by the Common Terminology Criteria for Adverse Events (CTCAE) v5.0.

SECONDARY OUTCOMES:
Rate of Reported Adverse Events Within 1 Month of Radiation | 1 Month
  The rate of reported adverse events (side effects) within 1 month of starting radiation as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Rate of Long-Term Adverse Events (Up to 2 Years) From the End of Radiation Rate of Long-Term Adverse Events (Up to 2 Years) From the End of Radiation | Up to 2 years after last dose of radiation
  The rates of reported long-term adverse events from the end of radiation up to a maximum of 2 years as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Overall Response Rate to Radiation Treatment | Up to 2 years after last dose of radiation
  Overall response rate to radiation (including irradiated and non-irradiated lesions) as assessed by computed tomography scans of lesions based on tumor measurements according to Response Evaluation Criteria in Solid Tumors (RECIST criteria Version 1.1 ).
Progression-Free Survival of Participants After Radiation Treatment | Up to 2 years after last dose of radiation
  Progression-free survival after radiation as assessed by computed tomography (CT) scans of lesions, tumor measurements according to Response Evaluation Criteria in Solid Tumors and clinical records.
Overall Survival After Radiation Treatment | Up to 2 years after last dose of radiation
  Overall survival after radiation as assessed by computed tomography (CT) scans of lesions, tumor measurements according to Response Evaluation Criteria in Solid Tumors(RECIST Version 1.1) and clinical records.
Local Control of Treated Lesions After Radiation Treatment | Up to 2 years after last dose of radiation
  Local control of the treated lesion as assessed by computed tomography (CT) scans of lesions, tumor measurements according to Response Evaluation Criteria in Solid Tumors (RECIST criteria Version 1.1 ) and clinical records.

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Hasan, MD, Principal Investigator — University of Chicago - Comprehensive Cancer Center
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF